CLINICAL TRIAL: NCT00005844
Title: A Phase I Study of Oxaliplatin in Children With Solid Tumors
Brief Title: Oxaliplatin in Treating Children With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067860; SJCRH-OXAL1 (Other: St. Jude Children's Research Hospital); NCI-T99-0059 (Other: National Cancer Institute)
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of oxaliplatin in treating children who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of oxaliplatin in children with advanced solid tumors.
* Determine the toxic effects of this drug in these patients.
* Determine the safety of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Assess the relationship between pharmacokinetic parameters and toxicity of this regimen and response in these patients.
* Determine the anti-tumor effects of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oxaliplatin IV over 2 hours on day 1 (every 3 weeks for up to 6 courses) OR on days 1, 14, and 28 (every 6 weeks for up to 3 courses). Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of oxaliplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Once the MTD for dose levels 1-4 is determined, an additional cohort of 3-6 patients is accrued and treated with oxaliplatin as above every 2 weeks (for up to 9 doses).

PROJECTED ACCRUAL: Approximately 6-20 patients will be accrued for this study within 1-3.3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic or unresectable solid tumors that are not amenable to standard treatment

  * Histological confirmation not required for brain stem tumors
* No known brain metastases
* No leukemia

PATIENT CHARACTERISTICS:

Age:

* 21 and under

Performance status:

* ECOG 0-2 OR
* Lansky 50-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3 (except with marrow involvement)
* Hemoglobin at least 8 g/dL
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin 0.2-1.4 mg/dL
* AST/ALT no greater than 3 times upper limit of normal

Renal:

* Creatinine normal for age OR
* Creatinine clearance at least 50 mL/min
* Electrolytes, calcium, and phosphorus normal

Cardiovascular:

* No symptomatic congestive heart failure, unstable angina, or cardiac arrhythmia

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No active graft-vs-host disease (GVHD)
* No allergy to platinum compounds or antiemetics
* No uncontrolled concurrent illness or infection
* No evidence of neuropathy
* Blood sugar normal

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 week since prior hematopoietic growth factors
* At least 3 months since prior stem cell transplantation and recovered

Chemotherapy:

* At least 3 weeks since prior chemotherapy (6 weeks for nitrosourea)

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 6 weeks since prior extensive radiotherapy to significant marrow-containing compartment
* At least 6 months since prior craniospinal radiotherapy; total abdominal, pelvic, or extensive lung radiotherapy; or mantle and Y-port radiotherapy
* At least 6 months since prior total body irradiation

Surgery:

* Not specified

Other:

* No concurrent therapy for GVHD
* No other concurrent anticancer investigational or commercial agents
* No other concurrent anticancer therapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2000-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheri L. Spunt, MD, Study Chair — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Result] Spunt SL, Freeman BB 3rd, Billups CA, McPherson V, Khan RB, Pratt CB, Stewart CF. Phase I clinical trial of oxaliplatin in children and adolescents with refractory solid tumors. J Clin Oncol. 2007 Jun 1;25(16):2274-80. doi: 10.1200/JCO.2006.08.2388. PMID 17538173
- [Result] Iacono LC, Spunt SL, Pratt CB, et al.: Pharmacokinetics of oxaliplatin in children with solid tumors. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-2170, 89b, 2002.
- [Result] Pratt CB, Spunt SL, Thompson SJ, et al.: Phase I Study of Oxaliplatin in Pediatric Patients with Malignant Solid Tumors. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-1498, 2001.
- See also: St. Jude Children's Research Hospital — http://stjude.org